CLINICAL TRIAL: NCT00555386
Title: A Pilot Study to Determine the Effect of Dietary Intervention on Novel Biomarkers of Breast Cancer Risk.
Brief Title: Soy, Selenium and Breast Cancer Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Quadram Institute Bioscience (Other); Big C Local Cancer Research and Care (Unknown); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Professor Aedin Cassidy, University of East Anglia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R14697; 07/Q0101/10
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Breast Cancer Risk
Keywords: Selenium; Soy; Breast Cancer Risk
MeSH Terms: interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): 6g of chocolate (supplemented with selenium and isoflavones) per day for the duration of one menstrual cycle (25-35 days)
  Interventions: Dietary Supplement: Soy and Selenium
- 2 (Placebo Comparator): 6g of chocolate (control) per day for the duration of one menstrual cycle (25-35 days)
  Interventions: Dietary Supplement: Soy and Selenium

INTERVENTIONS:
Dietary Supplement: Soy and Selenium — 6g of chocolate per day Control group with no supplementation Active group 50mg of soy protein isolate + 200µg selenium in the form of MSC

SUMMARY:
There is evidence to suggest that some dietary components can reduce the risk of breast cancer. In this pilot study two such components, isoflavones (compounds found in soy products) and selenium, will be given to women classed as at moderate to high risk of the disease. The aim is to determine some novel biomarkers of risk and to see the effect of supplementation on them.

DETAILED DESCRIPTION:
The high incidence of breast cancer, its relatively long development phase and the financial burden to the NHS in relation to treatment makes it a prime target for dietary preventative strategies. Epidemiological and experimental investigations suggest several key dietary components that may reduce breast cancer, in particular isoflavones and selenium. Few dietary intervention studies have been conducted to investigate putative protective effects, but with our growing understanding of cancer biology and the application of new -omics technologies it is now possible to use early biomarkers of risk to assess the potential efficacy of intervention studies.

In this pilot project, we will employ a combination of disciplines to examine the effect of dietary intervention in a group of women defined by NICE guidelines as being at increased risk (moderate-high) of developing breast cancer, using metabolomics to assess the tractability of biomarkers in response to the dietary intervention. Such trials are urgently needed to examine the protective effects of diet in women classified at increased risk and who are still in the 'zone of reversibility'. The results of this study will be used to justify and optimise larger scale intervention trials and ultimately to develop appropriate dietary recommendations for the prevention of breast cancer.

A dietary intervention study based on a randomised double-blind parallel design will be conducted in 30 pre-menopausal women (age 35-50) at moderate to high risk of developing breast cancer. The metabolomic profiles of urine and serum samples (collected at baseline and after dietary intervention) will be assessed. Participants will be randomised into two groups; the placebo group (consuming 6g of non-supplemented chocolate per day) and the supplemented group (consuming 6g of chocolate containing both soy and selenium per day). The intervention will last for the duration of one menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Pre menopausal women (age 35-50)at moderate to high risk of breast cancer based on family history (NICE guidelines)
* Attending Breast Clinic at NNUH
* Willing to consume 6g of chocolate per day for 25-35 days
* Regular menstrual cycle of 25-35 days in length

Exclusion Criteria:

* Current or previous diagnosis of breast cancer or cancer of any other site
* Diagnosis of hypertension (requiring active treatment)/diabetes/ coronary heart disease/ gastrointestinal disease/ any other systemic disease requiring treatment
* Regularly taking any prescribed medication within the last six months (including oral contraceptives)
* Fitted with a hormone releasing device
* Pregnant or lactating in the previous 12 months
* Using laxatives or antacids more than once a week
* Routinely taking soy or selenium supplements in the last twelve months
* Regularly taking any dietary or herbal supplements in the last six months
* Participation in any intervention study (soy or selenium) in the previous twelve months
* Parallel participation in another research study involving either dietary or medical intervention or sampling of biological fluids/materials
* Blood donation within sixteen weeks of study start/finish
* BMI <18.5 or >35
* Allergy to any chocolate/dairy/soy-based food products

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To determine the effect of supplementation with selenium and isoflavones on biomarkers of breast cancer risk. | 25-35 days

SECONDARY OUTCOMES:
Identify novel biomarkers of breast cancer risk through metabolomic analysis of samples collect. | 25-35 days

CONTACTS AND LOCATIONS:
Overall Officials: Aedin Cassidy, PhD, Principal Investigator — University of East Anglia
Locations (3):
- United Kingdom (3):
  - Institute of Food Research, Norwich, Norfolk
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - University of East Anglia, Norwich, Norfolk

REFERENCES:
- [Background] Akbaraly NT, Arnaud J, Hininger-Favier I, Gourlet V, Roussel AM, Berr C. Selenium and mortality in the elderly: results from the EVA study. Clin Chem. 2005 Nov;51(11):2117-23. doi: 10.1373/clinchem.2005.055301. Epub 2005 Aug 25. PMID 16123147
- [Background] Barnes S. Phytoestrogens and breast cancer. Baillieres Clin Endocrinol Metab. 1998 Dec;12(4):559-79. doi: 10.1016/s0950-351x(98)80004-9. PMID 10384813
- [Background] Bathen TF, Engan T, Krane J, Axelson D. Analysis and classification of proton NMR spectra of lipoprotein fractions from healthy volunteers and patients with cancer or CHD. Anticancer Res. 2000 Jul-Aug;20(4):2393-408. PMID 10953302
- [Background] Cassidy A, Bingham S, Setchell K. Biological effects of isoflavones in young women: importance of the chemical composition of soyabean products. Br J Nutr. 1995 Oct;74(4):587-601. doi: 10.1079/bjn19950160. PMID 7577895
- [Background] Cassidy A, Bingham S, Setchell KD. Biological effects of a diet of soy protein rich in isoflavones on the menstrual cycle of premenopausal women. Am J Clin Nutr. 1994 Sep;60(3):333-40. doi: 10.1093/ajcn/60.3.333. PMID 8074062
- [Background] Doll R, Peto R. The causes of cancer: quantitative estimates of avoidable risks of cancer in the United States today. J Natl Cancer Inst. 1981 Jun;66(6):1191-308. PMID 7017215
- [Background] Duncan AM, Merz BE, Xu X, Nagel TC, Phipps WR, Kurzer MS. Soy isoflavones exert modest hormonal effects in premenopausal women. J Clin Endocrinol Metab. 1999 Jan;84(1):192-7. doi: 10.1210/jcem.84.1.5387. PMID 9920082
- [Background] Duncan AM, Merz-Demlow BE, Xu X, Phipps WR, Kurzer MS. Premenopausal equol excretors show plasma hormone profiles associated with lowered risk of breast cancer. Cancer Epidemiol Biomarkers Prev. 2000 Jun;9(6):581-6. PMID 10868692
- [Background] El-Bayoumy K, Sinha R. Mechanisms of mammary cancer chemoprevention by organoselenium compounds. Mutat Res. 2004 Jul 13;551(1-2):181-97. doi: 10.1016/j.mrfmmm.2004.02.023. PMID 15225592
- [Background] Fan S, Meng Q, Auborn K, Carter T, Rosen EM. BRCA1 and BRCA2 as molecular targets for phytochemicals indole-3-carbinol and genistein in breast and prostate cancer cells. Br J Cancer. 2006 Feb 13;94(3):407-26. doi: 10.1038/sj.bjc.6602935. PMID 16434996
- [Background] Grover PL, Martin FL. The initiation of breast and prostate cancer. Carcinogenesis. 2002 Jul;23(7):1095-102. doi: 10.1093/carcin/23.7.1095. PMID 12117765
- [Background] Hu YJ, Diamond AM. Role of glutathione peroxidase 1 in breast cancer: loss of heterozygosity and allelic differences in the response to selenium. Cancer Res. 2003 Jun 15;63(12):3347-51. PMID 12810669
- [Background] Ip C. Lessons from basic research in selenium and cancer prevention. J Nutr. 1998 Nov;128(11):1845-54. doi: 10.1093/jn/128.11.1845. PMID 9808633
- [Background] Katdare M, Osborne M, Telang NT. Soy isoflavone genistein modulates cell cycle progression and induces apoptosis in HER-2/neu oncogene expressing human breast epithelial cells. Int J Oncol. 2002 Oct;21(4):809-15. PMID 12239620
- [Background] Lee SO, Nadiminty N, Wu XX, Lou W, Dong Y, Ip C, Onate SA, Gao AC. Selenium disrupts estrogen signaling by altering estrogen receptor expression and ligand binding in human breast cancer cells. Cancer Res. 2005 Apr 15;65(8):3487-92. doi: 10.1158/0008-5472.CAN-04-3267. PMID 15833885
- [Background] Li J, Orlandi R, White CN, Rosenzweig J, Zhao J, Seregni E, Morelli D, Yu Y, Meng XY, Zhang Z, Davidson NE, Fung ET, Chan DW. Independent validation of candidate breast cancer serum biomarkers identified by mass spectrometry. Clin Chem. 2005 Dec;51(12):2229-35. doi: 10.1373/clinchem.2005.052878. Epub 2005 Oct 13. PMID 16223889
- [Background] Lu J, Jiang C. Selenium and cancer chemoprevention: hypotheses integrating the actions of selenoproteins and selenium metabolites in epithelial and non-epithelial target cells. Antioxid Redox Signal. 2005 Nov-Dec;7(11-12):1715-27. doi: 10.1089/ars.2005.7.1715. PMID 16356132
- [Background] Messina MJ, Loprinzi CL. Soy for breast cancer survivors: a critical review of the literature. J Nutr. 2001 Nov;131(11 Suppl):3095S-108S. doi: 10.1093/jn/131.11.3095S. PMID 11694655
- [Background] Odunsi K, Wollman RM, Ambrosone CB, Hutson A, McCann SE, Tammela J, Geisler JP, Miller G, Sellers T, Cliby W, Qian F, Keitz B, Intengan M, Lele S, Alderfer JL. Detection of epithelial ovarian cancer using 1H-NMR-based metabonomics. Int J Cancer. 2005 Feb 20;113(5):782-8. doi: 10.1002/ijc.20651. PMID 15499633
- [Background] Paglia DE, Valentine WN. Studies on the quantitative and qualitative characterization of erythrocyte glutathione peroxidase. J Lab Clin Med. 1967 Jul;70(1):158-69. No abstract available. PMID 6066618
- [Background] Shah YM, Al-Dhaheri M, Dong Y, Ip C, Jones FE, Rowan BG. Selenium disrupts estrogen receptor (alpha) signaling and potentiates tamoxifen antagonism in endometrial cancer cells and tamoxifen-resistant breast cancer cells. Mol Cancer Ther. 2005 Aug;4(8):1239-49. doi: 10.1158/1535-7163.MCT-05-0046. PMID 16093440
- [Background] Rinaldi S, Peeters PH, Berrino F, Dossus L, Biessy C, Olsen A, Tjonneland A, Overvad K, Clavel-Chapelon F, Boutron-Ruault MC, Tehard B, Nagel G, Linseisen J, Boeing H, Lahmann PH, Trichopoulou A, Trichopoulos D, Koliva M, Palli D, Panico S, Tumino R, Sacerdote C, van Gils CH, van Noord P, Grobbee DE, Bueno-de-Mesquita HB, Gonzalez CA, Agudo A, Chirlaque MD, Barricarte A, Larranaga N, Quiros JR, Bingham S, Khaw KT, Key T, Allen NE, Lukanova A, Slimani N, Saracci R, Riboli E, Kaaks R. IGF-I, IGFBP-3 and breast cancer risk in women: The European Prospective Investigation into Cancer and Nutrition (EPIC). Endocr Relat Cancer. 2006 Jun;13(2):593-605. doi: 10.1677/erc.1.01150. PMID 16728585
- [Background] Solanky KS, Bailey NJ, Beckwith-Hall BM, Davis A, Bingham S, Holmes E, Nicholson JK, Cassidy A. Application of biofluid 1H nuclear magnetic resonance-based metabonomic techniques for the analysis of the biochemical effects of dietary isoflavones on human plasma profile. Anal Biochem. 2003 Dec 15;323(2):197-204. doi: 10.1016/j.ab.2003.08.028. PMID 14656525
- [Background] Solanky KS, Bailey NJ, Beckwith-Hall BM, Bingham S, Davis A, Holmes E, Nicholson JK, Cassidy A. Biofluid 1H NMR-based metabonomic techniques in nutrition research - metabolic effects of dietary isoflavones in humans. J Nutr Biochem. 2005 Apr;16(4):236-44. doi: 10.1016/j.jnutbio.2004.12.005. PMID 15808328
- [Background] Trock BJ, Hilakivi-Clarke L, Clarke R. Meta-analysis of soy intake and breast cancer risk. J Natl Cancer Inst. 2006 Apr 5;98(7):459-71. doi: 10.1093/jnci/djj102. PMID 16595782
- [Background] Tsubura A, Uehara N, Kiyozuka Y, Shikata N. Dietary factors modifying breast cancer risk and relation to time of intake. J Mammary Gland Biol Neoplasia. 2005 Jan;10(1):87-100. doi: 10.1007/s10911-005-2543-4. PMID 15886889
- [Background] Whanger PD. Selenium and its relationship to cancer: an update. Br J Nutr. 2004 Jan;91(1):11-28. doi: 10.1079/bjn20031015. PMID 14748935
- [Background] Xiang H, Schevzov G, Gunning P, Williams HM, Silink M. A comparative study of growth-inhibitory effects of isoflavones and their metabolites on human breast and prostate cancer cell lines. Nutr Cancer. 2002;42(2):224-32. doi: 10.1207/S15327914NC422_12. PMID 12416264
- [Background] Xu X, Duncan AM, Merz BE, Kurzer MS. Effects of soy isoflavones on estrogen and phytoestrogen metabolism in premenopausal women. Cancer Epidemiol Biomarkers Prev. 1998 Dec;7(12):1101-8. PMID 9865428
- [Background] Yang J, Xu G, Zheng Y, Kong H, Pang T, Lv S, Yang Q. Diagnosis of liver cancer using HPLC-based metabonomics avoiding false-positive result from hepatitis and hepatocirrhosis diseases. J Chromatogr B Analyt Technol Biomed Life Sci. 2004 Dec 25;813(1-2):59-65. doi: 10.1016/j.jchromb.2004.09.032. PMID 15556516
- [Background] Zhang J, Svehlikova V, Bao Y, Howie AF, Beckett GJ, Williamson G. Synergy between sulforaphane and selenium in the induction of thioredoxin reductase 1 requires both transcriptional and translational modulation. Carcinogenesis. 2003 Mar;24(3):497-503. doi: 10.1093/carcin/24.3.497. PMID 12663510
- [Background] Nutritional aspects of the development of cancer. Report of the Working Group on Diet and Cancer of the Committee on Medical Aspects of Food and Nutrition Policy. Rep Health Soc Subj (Lond). 1998;48:i-xiv, 1-274. No abstract available. PMID 9599404
- [Background] Clemons M, Goss P. Estrogen and the risk of breast cancer. N Engl J Med. 2001 Jan 25;344(4):276-85. doi: 10.1056/NEJM200101253440407. No abstract available. PMID 11172156